CLINICAL TRIAL: NCT04239716
Title: Feasibility of Combined Ultrasound Guided Interscalene Brachial Plexus Block and Erector Spinae Plane Block for Anesthesia in Modified Radical Mastectomy With Axillary Lymph Node Dissection: Pilot Study
Brief Title: Regional Anesthesia for Modified Radical Mastectomy With Axillary Lymph Node Dissection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Collaborators: Dr. Mohamed Elsayed Afandy (Unknown)
Responsible Party: Principal Investigator, Mona Raafat Elghamry, Dr. Mona Raafat Elghamry Assistant Professor of anesthesiology, Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: mastectomy regional anesthesia
Record Dates: First submitted 2020-01-18; First posted 2020-01-27 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Anesthesia, Conduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- regional anesthesia (Experimental): combination of erector spinae plane block (ESPB) and interscalene block(IB).the ESPB will be performed using linear ultrasound transducer (Philips® cx 50 extreme edition, USA) and we will inject 20 ml solution(10 ml 0.5% bupivacaine, 5 ml 2% lidocaine, and 5 ml normal saline). the IB will be performed using the same ultrasound machine and injecting the same solution
  Interventions: Other: regional anesthesia

INTERVENTIONS:
Other: regional anesthesia — combination of erector spinae plane block and interscalene block for anesthesia in modified radical mastectomy surgeries with axillary lymph node dissection

SUMMARY:
local and regional anesthesia have been introduced with the goal of reducing the side effects associated with general anesthesia and IV opioid analgesia.our hypothesis is that ultrasound-guided interscalene brachial plexus block and erector spinae plane block will provide efficient surgical anesthesia and postoperative analgesia after modified radical mastectomy.

DETAILED DESCRIPTION:
inadequate analgesia after modified radical mastectomy with axillary lymph node dissection may occur with most of regional anesthesia. pain in the axilla and upper limb is related to ineffective block of medial and lateral pectoral nerves as long thoracic and thoracodorsal nerves, leading to inadequate analgesia.The aim of this study is to evaluate the efficacy and safety of ultrasound-guided interscalene brachial plexus block and erector spinae plane block for providing surgical anesthesia and postoperative analgesia after modified radical mastectomy.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 40-85 years old
* American Society of Anesthesiologists' physical status III and IV
* Planned for modified radical mastectomy with axillary lymph node dissection

Exclusion Criteria:

* Patient refusal
* Neurological or psychiatric disorders
* Local infection at injection site
* Spine or chest wall deformity
* Allergy or any contraindication to any of the study drugs
* Opioid or alcoholic addiction
* Chronic pain of any cause
* Uncooperative patients.

Ages: 40 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Success rate of the regional blocks | from the start to the end of the operation
  completion of the surgery without need of general anesthesia.

SECONDARY OUTCOMES:
duration of the blocks | 24- hours in the postoperative period
  Time to first request of rescue analgesia postoperative
Patients' satisfaction | 24-hours postoperative
  degree of patients' satisfaction
Any adverse events | 24-hours postoperative
  postoperative nausea and vomiting, local anesthetic toxicity, desaturation, bradypnea,hypotension, bradycardia or somnolence

CONTACTS AND LOCATIONS:
Overall Officials: Mona R Elghamry, MD, Principal Investigator — Tanta University, Faculty of Medicine; Mohamed E Afandy, MD, Study Director — Tanta University, Faculty of Medicine
Locations (1):
- Tanta University, Faculty of Medicine, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Yes
statistics of the age ,BMI, duration of surgery,success rate, time of first analgesic request,patients' and surgeon's satisfaction, and complications
Supporting Information: SAP
Time Frame: Individual patient data will be shared after finishing and publication of the study.and it will be available for 1 year.
Access Criteria: the individual patient data will be available for scientific research only up on email request. request will be sent to email of principal investigator (drmonagh19802000@gmail.com)